CLINICAL TRIAL: NCT04110730
Title: The Influence of 3D Printed Prostheses on Neural Activation Patterns of the Primary Motor Cortex in Children With Unilateral Congenital Upper-limb Reductions
Brief Title: The Influence of 3D Printed Prostheses on Neural Activation Patterns
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0614-16-FB
Record Dates: First submitted 2019-09-22; First posted 2019-10-01 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Amniotic Band Syndrome; Upper Extremity Deformities, Congenital
MeSH Terms: conditions — Amniotic Band Syndrome; Upper Extremity Deformities, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 3D Prostheses Users (Experimental): Children with unilateral congenital upper-limb reductions
  Interventions: Device: 3D Printed Upper-limb Prosthesis; Behavioral: Home Intervention
- Typically Developing Children (Active Comparator): Age- and sex-matched control group of typically developing children.
  Interventions: Behavioral: Home Intervention

INTERVENTIONS:
Device: 3D Printed Upper-limb Prosthesis — The fingers and thumb were made of polylactic acid polymer manufactured using industrial 3D printers. The palm, socket, forearm brace, and leveraging structure were made of polylactic acid which has properties similar to thermoplastic that facilitate post manufacturing adjustments. Elastic cords placed inside the dorsal aspect of the fingers provided passive finger extension. Finger flexion was driven by non-elastic cords along the palmar surface of each finger and was activated through 20-30 degrees of wrist or elbow flexion.
  Other Names: Prosthesis use
  Arms: 3D Prostheses Users
Behavioral: Home Intervention — An occupational therapy student will perform 3 home visits a week and will direct a training protocol that consists of completing three trials of a series of 6 block building activities (i.e., block-stacking) for each hand separated by 30 seconds of rest (a total of 18 block building activities per hand). The block stacking activity consists in building a 4 block train, 3 cube bridge, 4 block wall, 3 block tower, 6 block steps, and 6 block pyramid. All subjects including the control group will perform the same home training protocol.
  Other Names: Block stacking activity

SUMMARY:
The neural basis underlying motor performance in children using a prosthesis has been severely understudied resulting in minimal empirical evidence. The use of functional near-infrared spectroscopy (fNIRS) in conjunction with customized and visually appealing 3D printed prostheses would provide the unique opportunity to quantitatively assess the influence of upper-limb prostheses in the neural activation patterns of the primary motor cortex and motor performance of children. This information would increase the investigators limited knowledge of how prosthesis usage influences the primary motor cortex of growing children and use this information to develop rehabilitation programs aimed at reducing prosthesis rejection and abandonment.

DETAILED DESCRIPTION:
The investigators anticipate enrolling a total of 40 children between 3 and 18 years of age. Specifically, two groups of children will be recruited; children with unilateral congenital upper-limb reductions (n=20) and age and sex-matched control group of typically developing children (n=20). Considering the effect size from preliminary data and to account for a 10% drop-out rate, a total sample of 40 subjects will provide 80% power to detect a true standardized effect size.

Participants will be asked to attend a total of 3 sessions. Participants will attend an initial measurement session to take a 3D scan of the affected and non-affected upper limbs as well as several anthropometric measurements. During this session, three pictures of the upper limbs will be taken which will also be used to verify the fit the prostheses in a process previously validated by our research team. The research participants will then be asked to come for two testing visits. During the first testing visit (visit 1), participants will be fitted with the prosthesis and required adjustments to improve comfort and avoid pressure point will be performed. After fitting the prosthesis, participants will be given 15 minutes to explore the prosthesis and adjust the tensioner dial to regulate the opening of the fingers to perform the Box and Block Test. After the training and accommodation period, participants will be asked to perform 3 trials of flexion and extension of each wrist with and without the prosthesis and 3 different trials of the Box and Blocks Test for each hand while monitoring neural activity of the primary motor cortex using a fNIRS device. After a period of 20 minutes rest, participants will be asked to perform three trials of a bimanual coordination test using an instrumented tray. The bimanual task will require participants to start from a standard position and then reach forward and grasp (hand-to-tray), transport and place a tray on a ledge (tray transport), and then return the hands to the starting position (hand return). This task will be performed unimanually (3 trials for each hand) and bimanually (3 trials using both hands). Eight weeks after the baseline measurements, participants will be asked to visit our laboratory for a second time and perform the same assessments. Between the testing visits, participants will be encouraged to use the prosthesis for a minimum of 2 hours a day. In addition, an occupational therapy student will perform 3 home visits a week and will direct a training protocol that consists of completing three trials of a series of 6 block building activities for each hand separated by 30 seconds of rest (a total of 18 block building activities per hand). All participants including the control group will perform the same training protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age 3-18 years.
* Individuals missing any digits, hand, arm, shoulder.
* Any dysfunction of the upper limbs.

Exclusion Criteria:

* Participants who are outside of age range.
* Participants with upper extremity injury within the past month.
* Medical conditions which would be contraindications to wear a prosthetic or assistive device, Such as skin abrasions and musculoskeletal injuries in the upper limbs.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change of mean values of brain hemodynamic responses | Change from baseline of mean values of brain hemodynamic responses at 8 weeks.
  The oxy-hemoglobin (HbO) and deoxy-hemoglobin (HbR) are two major chromospheres in the blood which absorb NIR light. The concentration of HbO and HbR varies in the capillary blood during the rest and task sessions. Thus, brain functional information can be revealed by the estimation of HbO and HbR. HbT is the total hemoglobin.
Change of hemispheric dominance | Change from baseline of hemispheric dominance at 8 weeks.
  Measured using the Laterality Index revealing hemispheric dominance. The Laterality index will reveal hemispheric dominance using the following formula:
  Laterality index=(Oxy l-Oxy r)/(Oxy l+Oxy r) In this equation, l represents the channels from the left hemisphere and r indicates the channels from the right hemisphere. The Laterality index value will reveal which channels in the group showed a higher change during the task. Positive values indicate left-hemisphere dominant activation, while negative values indicate a right-hemisphere dominant activation.
Change of synchrony of hand movement | Change from baseline of synchrony of hand movement at 8 weeks.
  The synchrony of hands movement will be quantified as the absolute temporal difference between hands (non-affected hand and affected hand with prosthesis) at six points in time while moving a bilateral instrumented tray.
Change of movement duration | Change from baseline of movement duration at 8 weeks.
  Movement duration for unimanual and bimanual tasks while using an instrumented tray.

SECONDARY OUTCOMES:
Satisfaction assessed by the Project-Prosthesis Satisfaction Inventory (CAPP-PSI). | after 8 weeks.
  The parents of the participants select a response for each question using the following categories which are scored from 0 to 4: "not at all" =0, "a little" =1, "somewhat" =2, "a lot" =3, or "very much" =4. A higher score indicates higher satisfaction. The CAPP-PSI is a standardized measure of prosthesis satisfaction in children with limb deficiency.
Satisfaction assessed by the Orthotics Prosthetics Users' Survey (OPUS). | after 8 weeks.
  The parents of the participants select a response for each question using the following categories which are scored from 5=Very Satisfied, 4= Somewhat satisfied, 3=Neither, satisfied nor dissatisfied, 2=Somewhat dissatisfied, 1=Very Dissatisfied. A higher score indicates higher satisfaction. The OPUS is a self-report questionnaire consisting of five modules. Module 5 (OPUS Satisfaction) will be used to assess different satisfaction element

CONTACTS AND LOCATIONS:
Overall Officials: Jorge M Zuniga, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska at Omaha, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
Unidentified data

REFERENCES:
- [Derived] Zuniga JM, Pierce JE, Copeland C, Cortes-Reyes C, Salazar D, Wang Y, Arun KM, Huppert T. Brain lateralization in children with upper-limb reduction deficiency. J Neuroeng Rehabil. 2021 Feb 3;18(1):24. doi: 10.1186/s12984-020-00803-1. PMID 33536034